CLINICAL TRIAL: NCT01551940
Title: Evaluation of Efficacy of Botulinum Toxin Type A in the Treatment of Sialorrhea in the Patient Affected by Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Toxin Treatment for Amyotrophic Lateral Sclerosis (ALS) Related Sialorrhea
Acronym: ALS-TOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010.607/11
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Sialorrhea; Amyotrophic Lateral Sclerosis
Keywords: Sialorrhea; Amyotrophic lateral sclerosis; Botulinum toxin
MeSH Terms: conditions — Sialorrhea; Amyotrophic Lateral Sclerosis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botox (Experimental): Botox injection : 100 UI of botulinum toxin type A (Botox®) diluted in 2.2 ml of NaCl 0.9 %
  Interventions: Drug: Botox injection
- Placebo (Placebo Comparator): Placebo injection : NaCl 0.9 %
  Interventions: Drug: Placebo injection

INTERVENTIONS:
Drug: Botox injection — Local ultrasound-guided bilateral injection of botulinum toxin type A in parotid (35 UI/gland) and submandibular (15 UI/gland) glands.
  Arms: Botox
Drug: Placebo injection — A local ultrasound-guided bilateral injection of placebo (NaCl 0.9 %) in parotid (0.7 ml/gland) and submandibular (0.3 ml/gland) glands.
  Arms: Placebo

SUMMARY:
Evaluation of the decrease of the secretion of saliva in patients with amyotrophic lateral sclerosis by a local ultrasound-guided bilateral injection of botulinum toxin type A in parotids and submandibular glands. The investigators want to demonstrate 1 month after the injection, by a multicenter French randomized double blind study, an improvement of at least 25 % of the functional embarrassment due to saliva, estimated with a visual analogue scale, a decrease of the quantity of saliva and a decrease of the embarrassment for the main caregiver.

DETAILED DESCRIPTION:
The patient will benefit from an ultrasound guided injection of botulinum toxin A (Botox®) or placebo (NaCl 0.9 %) and will be followed up in consultation at 4, 12, 16 (if reinjection) and 24 weeks. He will be contacted by telephone in 2 and in 8 weeks (percentage of decrease of functional embarrassment, percentage of decrease of salivary secretion rate). He can be able to benefit in the open label phase of a botulinum toxin type A injection at the 12-week follow up if he estimates that first injection was not effective or if the efficiency of the first injection began to become blurred. After the 6 months of the study, the patient will benefit again from the usual follow-up as advised by the French consensus conference in November, 2005.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Obtaining of a written consent after information
* Diagnosis of probable or certain ALS according to the El Escorial criteria of the World Federation and Neurology Committee on Neuromuscular Diseases
* Patient having a follow-up in an ALS center
* Sialorrhea with VAS functional embarrassment > or equal at 50/100.
* Patient beneficiary of Social Security regime

Exclusion Criteria:

* Evolving disease associated with predictable survival < 1 month
* Patient having previously received an injection of botulinum toxin in the salivary glands
* Patient taking the other medical treatments for sialorrhea in the 7 days before the inclusion in the study (scopoderm, trihexyph'nidyle, atropine, ipatropium, amitriptyline, clomipramine, oxybutinine, diphenhydramine, beta-blockers)
* Patient having benefited from radiotherapy or from surgery on the salivary glands
* Behavioral problems, dementia or other psychiatric problems
* Myasthenia
* Known Pregnancy or absence of contraception recognized as effective, breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Improvement of the functional embarrassment provoked by sialorrhea | 1 month after the injection
  Demonstrate after the injection of botulinum toxin type A an improvement of at least 25 % of the functional embarrassment provoked by sialorrhea in the ALS patient, evaluated with a horizontal visual analogue scale (VAS).

SECONDARY OUTCOMES:
Decrease of the salivary secretion rate and a decrease of the embarrassment for the main caregiver | 1 month after the injection
  Demonstrate, one month after the injection of botulinum toxin type A, a decrease of the salivary secretion rate and a decrease of the embarrassment for the main caregiver by a horizontal visual analogue scale.
Improvement of the value of the hypersalivation item in ALSFRS-R scale | 1 month after the injection
  Demonstrate, one month after the injection of botulinum toxin type A, an improvement of the value of the hypersalivation item in ALSFRS-R scale.
Decrease of the score of severity and frequency of the drooling rating scale | 1 month after the injection
  Demonstrate, one month after the injection of botulinum toxin type A, a decrease of the score of severity and frequency of the drooling rating scale
Decrease of the cotton roll weight | 1 month after the injection
  Demonstrate, one month after the injection of botulinum toxin type A, a decrease of the cotton roll weight.
  Cotton rolls weight: production and quantity of saliva are verified by placing dental cotton rolls during 3 minutes in the mouth of the patient and by comparing the weight of rolls dry and soaked with saliva.
Decrease of the number of paper handkerchiefs used | 1 month after the injection
  Demonstrate, one month after the injection of botulinum toxin type A, a decrease of the number of paper handkerchiefs used. We ask the patient to count the number of handkerchiefs used a day.
Modification of the speech evaluation | 1 month after the injection
  Demonstrate, one month after the injection of botulinum toxin typeA, a modification of the speech evaluation (evaluation realized by speech evaluator)
Improvement of the quality of life | 1 month after the injection
  Demonstrate, one month after the injection of botulinum toxin type A, an improvement of the quality of life. Scale to estimate quality of life (ALSAQ-40), usually used with the patients affected by ALS
Description of patient cohort after the first injection | 6 months after the injection
  Describe cohort after the first injection: evolution of scores for every patient among Day0 and Month1, delay of appearance of the efficiency, the duration of effect of the treatment, the side effects, the modification of the consistency of the saliva and the possible necessity for re-injecting the patient at 3 months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe VIAL, MD, Principal Investigator — Centre SLA, Groupement Hospitalier Est, Hôpital Neurologique Pierre Wertheimer, Hospices Civils de Lyon
Locations (13):
- France (13):
  - Département de Neurologie, Hôpital de l'Hôtel-Dieu, CHU d'Angers, Angers
  - Centre SLA, Groupement Hospitalier Est, Hôpital Neurologique Pierre Wertheimer, Hospices Civils de Lyon, Bron
  - Service de Neurologie Vastel, Hôpital Côte de Nacre, CHU de Caen, Caen
  - Service de Neurologie, Hôpital Gabriel Montpied, CHU de Clermont-Ferrand, Clermont-Ferrand
  - Centre SLA, Service de Neurologie A et pathologies du mouvement, Hôpital Roger Salengro, CHU de Lille, Lille
  - Service de Neurologie, Hôpital Dupuytren, CHU de Limoges, Limoges
  - Service de Neurologie, Hôpital de la Timone, CHU de Marseille, Marseille
  - Service de Neurologie, Hôpital Central, CHU de Nancy, Nancy
  - Centre de Référence maladies Neuromusculaires, Service de Médecine Physique et Réadaptation, Hôpital de l'Archet 1, CHU de Nice, Nice
  - Fédération des Maladies du Système Nerveux, Groupement Hospitalier Pitié Salpêtrière, AP-HP, Paris
  - Service de Neurologie, CHU de Saint-Etienne, Saint-Etienne
  - Département de Neurologie, Hôpital de Hautepierre, CHRU de Strasbourg, Strasbourg
  - Service d'Explorations Fonctionelles Neuro-Musculaires, Hôpital Rangueil, CHU de Toulouse, Toulouse